CLINICAL TRIAL: NCT00746733
Title: A Phase I, Open-Label, Randomized, Four Period Crossover Drug Interaction Study to Evaluate the Pharmacokinetic Profiles of VYVANSE™ and ADDERALL XR When Each is Administered Alone and in Combination With the Proton Pump Inhibitor Prilosec OTC™ in Healthy Adult Volunteers
Brief Title: Vyvanse and Adderall XR Given Alone and in Combination With Prilosec OTC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD489-113
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Drug; Interaction; Study
MeSH Terms: interventions — Lisdexamfetamine Dimesylate; SLI381

ARMS (2):
- Vyvanse (LDX) (Experimental)
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Adderall XR (AXR) (Experimental)
  Interventions: Drug: Adderall XR (mixed salts amphetamine)

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — 50mg capsule
  Arms: Vyvanse (LDX)
Drug: Adderall XR (mixed salts amphetamine) — 20mg capsule
  Arms: Adderall XR (AXR)

SUMMARY:
The purpose of this study is to determine if taking Vyvanse with Prilosec OTC or Adderall XR with Prilosec OTC changes how quickly the drug is absorbed into the body and/or changes how much of the drug is absorbed into the body.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, age 18 to 45 inclusive at the time of consent.
2. Male, or non-pregnant, non-lactating female
3. Female subjects must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening, and a negative urine pregnancy test on Day -1 after checking into the clinic the day before the first dose of investigational product.
4. Body Mass Index (BMI) between 20.0 and 30.0 kg/m² inclusive. This inclusion criterion will only be assessed at the first screening visit.
5. Satisfactory medical assessment with no significant or relevant abnormality in medical history, physical examination (PE), vital signs and laboratory evaluation
6. Normal or clinically insignificant Screening ECG findings as assessed by the Investigator.
7. Ability to swallow investigational products.

Exclusion Criteria:

1. Current or recurrent disease that could affect the action, absorption or disposition of the investigational products, or could affect clinical or laboratory assessments.
2. Current or relevant previous history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational products or study procedures.
3. Significant illness, as judged by the Investigator, within 2 weeks of the first dose of investigational product.
4. History of significant anxiety, tension or agitation as assessed by the Investigator.
5. History of or current diagnosis of glaucoma.
6. History of a seizure disorder (other than infantile febrile seizures), any tic disorder or a current diagnosis and/or known family history of Tourette's Disorder.
7. History of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
8. History of controlled or uncontrolled hypertension or a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg.
9. Known family history of sudden cardiac death or ventricular arrhythmia.
10. Currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently demonstrating suicidal ideation.
11. Current use of any medication (including prescription, over the counter [OTC], herbal or homeopathic preparations) with the exception of hormonal replacement therapy or hormonal contraceptives (Current use is defined as use within 14 days of first dose of investigational product).
12. Use of any medication known to inhibit or induce the CYP450 enzymes responsible for the metabolism of the investigational products within 14 days of first dose of investigational product.
13. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds or any of the stated ingredients.
14. History of alcohol or other substance abuse within the last year.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09-08 (Actual); Primary Completion 2008-10-26 (Actual); Study Completion 2008-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

REFERENCES:
- [Result] Haffey MB, Buckwalter M, Zhang P, Homolka R, Martin P, Lasseter KC, Ermer JC. Effects of omeprazole on the pharmacokinetic profiles of lisdexamfetamine dimesylate and extended-release mixed amphetamine salts in adults. Postgrad Med. 2009 Sep;121(5):11-9. doi: 10.3810/pgm.2009.09.2048. PMID 19820270
- [Derived] Wigal T, Brams M, Gasior M, Gao J, Giblin J. Effect size of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder. Postgrad Med. 2011 Mar;123(2):169-76. doi: 10.3810/pgm.2011.03.2275. PMID 21474905
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label, randomized, four period crossover
Groups:
- Vyvanse First: Vyvanse 50mg dosed once in the first intervention, Adderall XR 20 mg dosed once in the second intervention, Vyvanse 50mg + Prilosec OTC 40mg dosed once in the third intervention, Adderall XR 20mg + Prilosec OTC 40mg dosed once in the fourth intervention.
- Adderall XR First: Adderall XR 20 mg dosed once in the first intervention, Vyvanse 50mg dosed once in the second intervention, Adderall XR 20mg + Prilosec OTC 40mg dosed once in the third intervention, Vyvanse 50mg + Prilosec OTC 40mg dosed once in the fourth intervention.
Period: First Intervention
Arm/Group | Vyvanse First | Adderall XR First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Vyvanse First | Adderall XR First
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Third Intervention
Arm/Group | Vyvanse First | Adderall XR First
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Fourth Intervention
Arm/Group | Vyvanse First | Adderall XR First
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of d-Amphetamine for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Description: d-Amphetamine is an isomer of Vyvanse and Adderall XR and is an active form that is responsible for the drug's therapeutic activity.
Time Frame: 0 through 96 hours after dosing
Population: Pharmacokinetic (PK) population defined as all subjects who have evaluable concentration-time profiles.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
ng/ml | 45.04 (13.971) | 28.66 (7.174) | 46.34 (9.710) | 29.97 (5.719)

2. Secondary Outcome: Drug Rating Questionnaire-Subject (DRQ-S), Question 2, for Vyvanse and Adderall XR in Combination With Prilosec OTC.
Description: Question 2: How much do you like the effects you are feeling now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12 and 24 hours after dosing
Population: Pharmacodynamic (PD) population defined as all subjects who have evaluable DRQ-S values reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 21 | 21
units on a scale
  Pre-dose | 1.0 (0.0) | 1.0 (0.0)
  0.5 h | 1.2 (0.60) | 2.0 (3.09)
  1 h | 1.8 (1.75) | 2.0 (3.08)
  1.5 h | 4.6 (8.28) | 2.2 (3.56)
  2 h | 4.6 (8.33) | 2.5 (4.56)
  2.5 h | 3.9 (6.04) | 2.3 (3.73)
  3 h | 3.5 (5.78) | 1.5 (1.03)
  3.5 h | 2.7 (3.78) | 1.3 (0.80)
  4 h | 1.7 (1.06) | 1.4 (0.86)
  5 h | 2.4 (3.93) | 1.3 (0.72)
  6 h | 1.4 (0.81) | 1.2 (0.51)
  8 h | 1.4 (0.74) | 1.3 (1.32)
  12 h | 1.2 (0.62) | 1.1 (0.36)
  24 h | 1.3 (0.72) | 1.0 (0.22)

3. Secondary Outcome: DRQ-S, Question 1, for Vyvanse and Adderall XR in Combination With Prilosec OTC
Description: Question 1: How much do you feel the drug now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12 and 24 hours after dosing
Population: PD population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 21 | 21
units on a scale
  Pre-dose | 1.0 (0.0) | 1.0 (0.0)
  0.5 h | 1.3 (0.73) | 1.3 (0.66)
  1 h | 2.1 (2.66) | 1.9 (2.46)
  1.5 h | 5.2 (8.38) | 2.3 (2.97)
  2 h | 6.0 (8.69) | 3.5 (5.33)
  2.5 h | 6.0 (7.59) | 3.5 (4.64)
  3 h | 5.3 (6.72) | 2.7 (3.36)
  3.5 h | 4.9 (6.09) | 2.1 (2.01)
  4 h | 3.8 (4.57) | 2.1 (1.84)
  5 h | 3.1 (4.13) | 1.9 (1.74)
  6 h | 3.4 (3.60) | 1.5 (0.87)
  8 h | 3.0 (4.26) | 1.3 (0.66)
  12 h | 4.4 (7.19) | 1.2 (0.54)
  24 h | 1.6 (1.40) | 1.0 (0.22)

4. Secondary Outcome: DRQ-S, Question 3, for Vyvanse and Adderall XR in Combination With Prilosec OTC
Description: Question 3: Do you dislike the drug effect you are feeling now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12 and 24 hours after dosing
Population: PD population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 21 | 21
units on a scale
  Pre-dose | 1.0 (0.0) | 1.0 (0.0)
  0.5 h | 2.0 (3.49) | 2.1 (3.11)
  1 h | 1.8 (1.67) | 2.0 (3.08)
  1.5 h | 4.3 (8.03) | 1.8 (1.55)
  2 h | 4.5 (8.37) | 1.4 (0.93)
  2.5 h | 3.8 (6.39) | 1.4 (0.80)
  3 h | 3.4 (5.78) | 1.2 (0.54)
  3.5 h | 2.6 (3.54) | 1.3 (0.72)
  4 h | 1.8 (1.18) | 1.3 (0.80)
  5 h | 2.3 (4.13) | 1.3 (0.97)
  6 h | 1.6 (1.02) | 1.2 (0.70)
  8 h | 1.6 (1.78) | 1.1 (0.48)
  12 h | 1.3 (0.80) | 1.2 (0.51)
  24 h | 1.1 (0.48) | 1.0 (0.22)

5. Secondary Outcome: Systolic Blood Pressure for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Time Frame: Pre-dose and 1, 2, 4, 8, 12, 24, 48, 72 and 96 hours after dosing
Population: Safety population defined as subjects who take at least one dose of investigational medicinal product and have at least one post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
mmHg
  Pre-dose | 115.6 (10.79) | 115.3 (10.26) | 114.8 (11.29) | 113.9 (11.71)
  1 h | 122.8 (11.10) | 121.0 (10.46) | 121.7 (13.31) | 122.6 (9.67)
  2 h | 127.9 (12.81) | 122.2 (11.34) | 125.5 (10.14) | 124.7 (12.74)
  4 h | 127.6 (12.95) | 120.8 (11.71) | 125.2 (11.50) | 124.2 (9.75)
  8 h | 126.0 (12.69) | 122.4 (11.04) | 123.5 (13.25) | 119.2 (10.99)
  12 h | 123.4 (15.62) | 121.9 (12.04) | 122.2 (13.19) | 118.4 (10.58)
  24 h | 114.0 (11.68) | 118.1 (12.97) | 114.7 (11.19) | 115.6 (13.42)
  48 h | 114.6 (12.84) | 112.6 (10.56) | 114.4 (10.81) | 113.6 (11.01)
  72 h | 113.7 (10.25) | 114.8 (11.81) | 115.1 (11.71) | 116.0 (9.74)
  96 h | 114.0 (10.53) | 114.5 (10.72) | 114.8 (11.06) | 116.1 (9.29)

6. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of d-Amphetamine for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Description: as for outcome 1
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
h | 3.5 (1.14) | 5.2 (3.10) | 3.5 (0.97) | 3.3 (1.45)

7. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of d-Amphetamine for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Description: as for outcome 1
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
ng.h/ml | 626.27 (198.982) | 473.70 (71.043) | 687.00 (196.906) | 472.35 (108.891)

8. Primary Outcome: Terminal Half-life (T 1/2) of d-Amphetamine for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Description: as for outcome 1
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
h | 9.7 (1.55) | 10.25 (1.36) | 10.4 (1.65) | 10.91 (1.95)

9. Secondary Outcome: Diastolic Blood Pressure for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Time Frame: Pre-dose and 1, 2, 4, 8, 12, 24, 48, 72 and 96 hours after dosing
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
mmHg
  Pre-dose | 76.0 (6.68) | 74.1 (6.72) | 77.7 (8.60) | 75.8 (7.80)
  1 h | 79.2 (6.62) | 76.4 (5.98) | 80.5 (9.52) | 80.4 (6.29)
  2 h | 79.0 (6.97) | 75.4 (6.58) | 82.0 (6.44) | 81.9 (8.71)
  4 h | 79.9 (7.91) | 77.7 (6.31) | 82.0 (7.68) | 82.0 (7.09)
  8 h | 78.6 (7.87) | 74.1 (5.73) | 80.3 (9.54) | 79.2 (7.96)
  12 h | 79.6 (9.45) | 78.5 (8.29) | 78.7 (10.47) | 77.8 (8.20)
  24 h | 75.9 (6.76) | 76.8 (8.62) | 75.0 (7.76) | 75.4 (7.30)
  48 h | 74.5 (8.39) | 73.5 (8.40) | 77.2 (6.53) | 74.4 (8.01)
  72 h | 75.1 (7.97) | 74.7 (7.24) | 76.1 (7.58) | 77.9 (6.77)
  96 h | 74.5 (8.02) | 75.7 (7.65) | 75.7 (7.48) | 78.3 (6.96)

10. Secondary Outcome: Pulse Rate for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Time Frame: Pre-dose and 1, 2, 4, 8, 12, 24, 48, 72 and 96 hours after dosing
Population: Safety population
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
bpm
  Pre-dose | 70.9 (9.87) | 69.0 (8.87) | 73.3 (10.16) | 71.4 (10.14)
  1 h | 69.7 (10.61) | 70.0 (11.29) | 73.4 (10.91) | 73.8 (13.78)
  2 h | 78.2 (11.64) | 75.2 (10.85) | 83.4 (14.68) | 80.5 (16.87)
  4 h | 79.0 (14.40) | 74.5 (12.62) | 84.4 (16.29) | 78.4 (15.03)
  8 h | 84.8 (11.38) | 79.1 (10.70) | 87.7 (14.34) | 81.5 (11.50)
  12 h | 86.4 (13.84) | 82.3 (14.12) | 89.1 (13.77) | 82.7 (10.99)
  24 h | 79.9 (11.19) | 74.7 (12.58) | 80.4 (11.32) | 76.4 (12.06)
  48 h | 73.2 (11.28) | 74.0 (11.02) | 75.1 (10.32) | 75.0 (9.46)
  72 h | 72.2 (10.63) | 73.3 (9.16) | 72.0 (7.99) | 72.7 (8.78)
  96 h | 70.7 (10.64) | 70.4 (9.11) | 72.5 (10.12) | 73.9 (9.86)

11. Secondary Outcome: Electrocardiogram Results (QTcF Interval) for Vyvanse and Adderall XR Alone and in Combination With Prilosec OTC
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate(e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Pre-dose, 2 and 8 hours after dosing
Population: Safety population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 24 | 23 | 21 | 21
msec
  Pre-dose | 399.8 (14.55) | 398.3 (15.24) | 399.3 (13.38) | 399.8 (15.04)
  2 h | 395.0 (14.11) | 394.6 (13.42) | 397.9 (13.86) | 396.1 (14.49)
  8 h | 390.0 (12.45) | 393.8 (13.94) | 395.4 (14.93) | 394.4 (13.26)

12. Primary Outcome: Cmax of l-Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: l-Amphetamine is an isomer of Adderall XR and is an active form that is responsible for the drug's therapeutic activity.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
ng/ml | 7.91 (2.022) | 8.10 (1.632)

13. Primary Outcome: Tmax of l-Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: l-Amphetamine is an isomer of Adderall XR and is an active form that is responsible for the drug's therapeutic activity.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
h | 5.6 (3.0) | 3.5 (1.74)

14. Primary Outcome: AUC of l-Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
ng.h/ml | 145.28 (24.355) | 145.83 (38.233)

15. Primary Outcome: T 1/2 of l-Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: l-Amphetamine is an isomer of Adderall XR and is an active form that is responsible for the drug's therapeutic activity.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
h | 11.98 (1.92) | 13.06 (2.63)

16. Primary Outcome: Cmax of Total Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: Total amphetamine is the d- and l-amphetamines.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
ng/ml | 36.56 (9.188) | 38.05 (7.351)

17. Primary Outcome: Tmax of Total Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: Total amphetamine is the d- and l-amphetamines.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
h | 5.30 (3.07) | 3.29 (1.45)

18. Primary Outcome: AUC of Total Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: Total amphetamine is the d- and l-amphetamines.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
ng.h/ml | 620.68 (95.689) | 620.91 (145.378)

19. Primary Outcome: T 1/2 of Total Amphetamine for Adderall XR Alone and in Combination With Prilosec OTC
Description: Total amphetamine is the d- and l-amphetamines.
Time Frame: 0 through 96 hours after dosing
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Adderall XR | Adderall XR + Prilosec OTC
Number analyzed (Participants) | 23 | 21
h | 10.38 (1.56) | 11.05 (2.22)

ADVERSE EVENTS:
Arm/Group | Vyvanse | Adderall XR | Vyvanse + Prilosec OTC | Adderall XR + Prilosec OTC
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 8/24 | 3/23 | 10/21 | 3/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vyvanse (N=24) | Adderall XR (N=23) | Vyvanse + Prilosec OTC (N=21) | Adderall XR + Prilosec OTC (N=21)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 8 (9) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.